CLINICAL TRIAL: NCT02933372
Title: Cholinergic Mechanisms of Gait Dysfunction in Parkinson's Disease Experiments 1 & 2 - Projects #3
Brief Title: Cholinergic Mechanisms of Gait Dysfunction in Parkinson's Disease Experiments 1 & 2 - Proj #3
Acronym: UdallP3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roger L. Albin, Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00093188
Record Dates: First submitted 2016-04-06; First posted 2016-10-14 (Estimated); Results first posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: All participants (Parkinson's disease patients and healthy controls) will receive the study drug varenicline.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Parkinson's Disease Patients (Experimental): Participants take varenicline for several days and have two Positron Emission Tomography (PET) scans. PET scans are used to estimate how much varenicline is actually in the brain. Safety monitoring with clinical assessments of severity of Parkinson disease (PD) and cognition are performed.
  Interventions: Drug: Varenicline
- Healthy Controls (Experimental): Participants take varenicline for several days and have two Positron Emission Tomography (PET) scans. The PET scans are used to estimate how much varenicline is actually in the brain. Safety monitoring with clinical assessments for presence of Parkinson disease (PD) and cognition are performed.
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Participants take varenicline for 10 days. Each participant will be on one dosage throughout the 10 days, but not all participants receive the same dosage. The dosages that were utilized for both Parkinson's disease participants and healthy volunteers were 0.25mg once a day, 0.25mg twice a day, and 0.5mg twice a day. A fourth dosing group of 1 mg varenicline twice a day was studied in Parkinson's disease participants, but not in healthy volunteers.
  Other Names: Chantix

SUMMARY:
Varying oral doses of Varenicline (VCN), starting with very low doses, will be administered to participants with Parkinson's Disease (PD) or healthy controls without PD for several days. Positron emission tomography (PET) scans after administration of VCN will be used to determine the lowest oral dose of VCN producing an adequate brain level of VCN. These experiments (1 & 2) will be used to determine an appropriate oral dose of VCN to administer to PD participants for experiment 3 of the study (see NCT04403399).

DETAILED DESCRIPTION:
To demonstrate that α4β2* nAChRs are appropriate therapeutic targets in Parkinson's Disease (PD), it is necessary to study key pharmacokinetic-pharmacodynamic features of α4β2* nAChR in the context of the PD brain with loss of nerve cells that produce the neurotransmitter acetylcholine, a pathologic environment in which they may exhibit unique features. This personalized medicine approach focuses our studies on the subgroup of PD subjects with loss of nerve cells that produce the neurotransmitter acetylcholine identified by Project II and the Clinical Resource Core. The investigators will assess α4β2* nAChR features using PET imaging with the α4β2* nAChR ligand [18 - Fluorine] flubatine, subacute administration of the α4β2* nAChR partial agonist Varenicline (VCN), and laboratory measures of gait, balance, and attention. The investigators will use [18 - Fluorine] flubatine PET to assess VCN occupancy of brain α4β2* nAChRs (experiments 1 & 2). VCN will be administered to both PD participants (experiment 1) and healthy controls (experiment 2) and both populations will undergo a flubatine PET scan to assess VCN occupancy. Using this PET data to select an appropriate VCN dose, the investigators will perform a pharmacodynamic study (experiment 3) with subacute VCN administration to determine if α4β2* nAChR stimulation improves laboratory measures of gait function, postural control, and attentional function in PD subjects with loss of nerve cells that produce the neurotransmitter acetylcholine.

ELIGIBILITY:
Inclusion Criteria:

1. PD diagnosis will be based on the United Kingdom Parkinson's Disease Society Brain Bank Research Center (UKPDSBRC) clinical diagnostic criteria. The investigators will enrich the cohort by recruiting subjects at modified Hoehn and Yahr stages 2 or higher, duration of motor disease 5 years or longer, age >65 years, or the Postural Instability and Gait Disorder (PIGD) phenotype. Duration of motor disease will be defined as the time between onset of motor symptoms and time of entry into the study. The PIGD phenotype is defined as described previously. PD subjects with defined cholinergic deficits will be recruited as described in Project II. PD subjects will have cortical cholinergic deficits based on 5th percentile cutoff of the normal controls as defined previously.
2. Stable dopaminergic replacement therapy for 3 months prior to enrollment and expected to maintain stable dopaminergic therapy for duration of study participation.

Exclusion Criteria:

1. Other disorders which may resemble PD with or without dementia, such as vascular dementia, normal pressure hydrocephalus, progressive supranuclear palsy, multiple system atrophy, corticobasal ganglionic degeneration, or toxic causes of parkinsonism. Prototypical cases have distinctive clinical profiles, like vertical supranuclear gaze palsy, early and severe dysautonomia or appendicular apraxia, which may differentiate them from idiopathic PD. The use of the UKPDSBRC clinical diagnostic criteria for PD will mitigate the inclusion of subjects with atypical parkinsonism and all participants will undergo [11-Carbon]dihydrotetrabenazine PET to confirm striatal dopaminergic denervation.
2. Subjects on neuroleptic, anticholinergic (trihexphenidyl, benztropine), or cholinesterase inhibitor drugs.
3. Current or previous (within last 6 months) use of any product or medication containing nicotinic agents,including use of tobacco products such as cigarettes, cigars, pipes, chewing tobacco, etc., electronic cigarettes, over-the-counter nicotine patches, chewing gum containing nicotine, or varenicline.
4. Evidence of a stroke or mass lesion on structural brain imaging (MRI).
5. Participants in whom magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.
6. Severe claustrophobia precluding MR or PET imaging
7. Subjects limited by participation in research procedures involving ionizing radiation.
8. Pregnancy (test within 48 hours of each PET session) or breastfeeding.
9. Significant risk of cardiovascular event.
10. Active, significant mood disorder.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Albin, MD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Parkinson's Disease Patients: Participants take varenicline for 10 days. Each participant will be on one dosage throughout the 10 days, but not all participants receive the same dosage. The dosages that were utilized were 0.25mg once a day, 0.25mg twice a day, 0.5mg twice a day and 1mg twice a day.
- Healthy Controls: Participants take varenicline for 10 days. Each participant will be on one dosage throughout the 10 days, but not all participants receive the same dosage. The dosages that were utilized were 0.25mg once a day, 0.25mg twice a day, and 0.5mg twice a day.
Period: Overall Study
Arm/Group | Parkinson's Disease Patients | Healthy Controls
Started | 15 | 10
Completed | 15 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All consented participants
Groups:
- Healthy Controls: : Participants take varenicline for 10 days. Each participant will be on one dosage throughout the 10 days, but not all participants receive the same dosage. The dosages that were utilized were 0.25mg once a day, 0.25mg twice a day, and 0.5mg twice a day.
- Total: Total of all reporting groups
Arm/Group | Parkinson's Disease Patients | Healthy Controls | Total
Number analyzed (Participants) | 15 | 10 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (5.20) | 66.4 (8.95) | 66.9 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 14 | 8 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 10 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 10 | 25
MDS-UPDRS III [Mean (Standard Deviation); unit: units on a scale] — Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III (motor examination) includes 18 items (33 scores). Each item scores from 0 (normal) to 4 (severe) and total score is obtained from the sum of the corresponding item scores. The minimum is 0, maximum is 132, with higher scores indicating more disability.
  units on a scale | 31.9 (12.83) | 3.5 (1.84) | 20.5 (17.27)
Geriatric Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Geriatric Depression Scale (GDS) is a 30-item questionnaire (long form) to measure depression in the older population. Participants are asked to respond yes or no to how they felt over the past week. Scores range from 0 to 30, with higher scores indicating more severe depression.
  units on a scale | 3.2 (3.75) | 1.6 (2.01) | 2.6 (3.22)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — Montreal Cognitive Assessment (MoCA) is a questionnaire assessing cognitive dysfunction. It assesses attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The score ranges from 0 to 30, with lower scores indicating more severe cognitive impairment.
  units on a scale | 25.5 (1.73) | 26.8 (2.30) | 26.0 (2.04)

OUTCOME MEASURES:

1. Primary Outcome: Varenicline Occupancy of alpha4beta2* Nicotinic Acetylcholine Receptors
Description: Varenicline occupancy of alpha4beta2* nicotinic acetylcholine receptors (nAChR) was assessed with ascending doses of varenicline and the selective alpha4beta2* nAChR positron emission tomography (PET) ligand [18F]Flubatine. Alpha4beta2* nAChR agonists may induce nAChR expression. Consequently, we imaged participants at the end of their drug exposure periods (Day 10) and again after 5 days (~5 half-lives) of washout from drug exposure (Day 15). We used the difference between the two PET scans, (Day 10 - Day 15)/Day 15 x 100%, to determine the receptor occupancy of alpha4beta2* nicotinic acetylcholine receptors (nAChR) by each dose of varenicline.
Time Frame: 15 days
Population: All consented and treated participants who had adequate PET scans. In Parkinson's Disease cohort, there were technical difficulties with PET scans in 5 participants. In the Healthy Controls cohort, one participant's data was excluded because of suspected covert tobacco abuse and there were technical difficulties with the PET scan for one participant.
Measure: Mean (Standard Deviation); unit: percentage of VCN-alpha4beta2* nAChRs
Groups:
- Parkinson's Disease Patients: Participants take varenicline for several days and have two Positron Emission Tomography (PET) scans. PET scans are used to estimate how much varenicline is actually in the brain. Safety monitoring with clinical assessments of severity of Parkinson disease (PD) and cognition are performed.
  Varenicline: Participants take varenicline for 10 days. Each participant will be on one dosage throughout the 10 days, but not all participants receive the same dosage. The dosages that were utilized were 0.25mg once a day, 0.25mg twice a day, 0.5mg twice a day and 1mg twice a day.
  [18-Fluorine] Flubatine PET Scan: Participants will undergo 2 different PET scanning sessions. Radiotracers will be injected into the participant's vein through an IV (intravenous catheter or plastic "tube" inserted in an arm vein). A tracer refers to a small amount of a radioactive substance that does not alter body function.
  Evaluation by Investigator: Participants will undergo cognitive testing, a physical exam, and gait and posture assessments
- Healthy Controls: Participants take varenicline for several days and have two Positron Emission Tomography (PET) scans. The PET scans are used to estimate how much varenicline is actually in the brain. Safety monitoring with clinical assessments for presence of Parkinson disease (PD) and cognition are performed.
  Varenicline: Participants take varenicline for 10 days. Each participant will be on one dosage throughout the 10 days, but not all participants receive the same dosage. The dosages that were utilized were 0.25mg once a day, 0.25mg twice a day, 0.5mg twice a day and 1mg twice a day.
  [18-Fluorine] Flubatine PET Scan: Participants will undergo 2 different PET scanning sessions. Radiotracers will be injected into the participant's vein through an IV (intravenous catheter or plastic "tube" inserted in an arm vein). A tracer refers to a small amount of a radioactive substance that does not alter body function.
  Evaluation by Investigator: Participants will undergo cognitive testing, a physical exam, and gait and posture assessments
Arm/Group | Parkinson's Disease Patients | Healthy Controls
Number analyzed (Participants) | 10 | 9
percentage of VCN-alpha4beta2* nAChRs
  0.25 mg once daily Varenicline: number analyzed (Participants) | 2 | 3
  0.25 mg once daily Varenicline | 67.0 (4.9) | 67.9 (3.1)
  0.25 mg twice daily Varenicline: number analyzed (Participants) | 3 | 3
  0.25 mg twice daily Varenicline | 65.7 (8.0) | 70.6 (1.9)
  0.5 mg twice daily Varenicline: number analyzed (Participants) | 3 | 3
  0.5 mg twice daily Varenicline | 66.3 (5.0) | 69.6 (4.0)
  1 mg twice daily Varenicline: number analyzed (Participants) | 2 | 0
  1 mg twice daily Varenicline | 71.5 (10.6) |

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Parkinson's Disease Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/10
Other Adverse Events (participants affected / at risk) | 6/15 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parkinson's Disease Patients (N=15) | Healthy Controls (N=10)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stomach cramping (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood in urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Tiredness (General disorders) | 1 (1) | 0 (0)
ended PET scan prior to completion (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT02933372/SAP_000.pdf
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT02933372/Prot_001.pdf